CLINICAL TRIAL: NCT04220762
Title: A Clinical Study to Determine the Optimal Dose of WIN-1001X by Evaluating Its Efficacy and Safety in Patients With Early Parkinson's Disease: Double-blind, Randomized, Placebo-controlled, Multicenter, Phase II Study
Brief Title: A Study to Determine the Dose of WIN-1001X by Evaluating Efficacy and Safety in Early Parkinson's Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medi Help Line (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIN-1001X-P2
Record Dates: First submitted 2019-12-17; First posted 2020-01-07 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group 1 (Experimental): The randomized patients are administered 3 tablets of the investigational product (400mg) twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Interventions: Drug: WIN-1001X
- Test Group 2 (Experimental): The randomized patients are administered 3 tablets of the investigational product (800mg) twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Interventions: Drug: WIN-1001X
- Test Group 3 (Experimental): The randomized patients are administered 3 tablets of the investigational product (1200mg) twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Interventions: Drug: WIN-1001X
- Placebo group (Placebo Comparator): The randomized patients are administered 3 tablets of the placebo drug twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WIN-1001X — This study has been designed as a randomized, double-blind, and placebo-controlled study.
  Once the patients who have voluntarily singed an informed consent form are enrolled in this study, their eligibilities for the study are assessed and those who have satisfied the inclusion/exclusion criteria are randomized to the test group 1 (400mg), 2 (800mg), and 3 (1200mg), or the control group (placebo group) in a ratio of 1:1:1:1. The randomized patients are administered 3 tablets of the investigational product twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Arms: Test Group 1; Test Group 2; Test Group 3
Drug: Placebo — This study has been designed as a randomized, double-blind, and placebo-controlled study.
  Once the patients who have voluntarily singed an informed consent form are enrolled in this study, their eligibilities for the study are assessed and those who have satisfied the inclusion/exclusion criteria are randomized to the test group 1 (400mg), 2 (800mg), and 3 (1200mg), or the control group (placebo group) in a ratio of 1:1:1:1. The randomized patients are administered 3 tablets of the investigational product twice a day for 12 weeks and the safety follow-up should be carried out for 2 weeks after administration of the investigational product is terminated.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine the optimal dose of WIN-1001X for its therapeutic confirmatory study by comparing and evaluating the efficacy and safety of each dose group by conducting a therapeutic exploratory study on three dose groups of WIN-1001X 400 mg, 800 mg, and 1200 mg, and placebo group in patients with early Parkinson's disease.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the difference in the change of MDS UPDRS Part Ⅲ between WIN-1001X 400 mg, 800 mg, and 1200 mg as the test drugs compared to placebo as the control drug after administering them for 12 weeks.

The secondary objectives of this study are to evaluate the therapeutic efficacy and safety of the 3 dose groups of WIN-1001X compared to placebo group by assessing the changes in MDS UPDRS Part Ⅲ after administering the investigational products for 4 and 8 weeks, the changes in MDS UPDRS Part Ⅰ, Part Ⅱ, Part Ⅰ+Part Ⅱ+Part Ⅲ, and Modified Hoehn and Yahr scale after administering for 4, 8, and 12 weeks, the changes in K-NMSS (Non-Motor Symptoms Scale), K-MoCA (Korean-Montreal Cognitive Assessment), K-PDQ-39 (Parkinson's Disease Questionnaire) score.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥30 years old at the time of informed consent
* Subjects diagnosed with Parkinson's disease satisfying the UKPDSBB (United Kingdom Parkinson's Disease Society Brain Bank) Clinical Diagnostic Criteria and showing decreased dopamine transporters in the dopamine transporter imaging (e.g.: ¹⁸F-FP-CIT PET, etc.)
* Modified Hoehn and Yahr stage ≤ 3.0
* K-MMSE (Korean Mini-Mental State Examination) score ≥20 at the screening visit (visit 1)
* Subjects who can understand and follow the instructions on this clinical study, and fully participate in the clinical study
* MDS UPDRS Part Ⅱ+Part Ⅲ score ≥18 at baseline (visit 2)
* Subjects who have voluntarily determined to participate in this study and signed the written informed consent form

Exclusion Criteria:

* Atypical or secondary parkinsonism or benign tremulous parkinsonism
* History of treatments with levodopa, dopamine agonists, anticholinergics, MAO-B inhibitors, COMT inhibitors, amantadine, or NMDA receptor antagonists (However, subjects who have not been administered such drugs for at least 6 months in a row and have no history of treatment within 4 weeks prior to their written consent can be enrolled)
* In case the investigators determine the symptom control is difficult with placebo
* Hypersensitivity to herbal medicine
* Subjects with dementia whose K-MMSE score is ≤19, severe psychopathy requiring treatment or hallucination
* Any disorder that may affect the absorption, distribution, metabolism, and excretion of drugs
* History of surgical treatment for Parkinson's disease
* Subjects who have been administered another investigational product within 30 days prior to screening
* Female subjects who are pregnant or lactating, or who have child-bearing potential (i.e., (i) those who are not surgically non-infertile, or (ii) who are not using adequate contraceptive methods [including at least one of the barrier methods], or (iii) who are not sexually abstinent, or (iv) for whom at least 2 years have not elapsed since their last menstruation)
* History of chronic alcohol or drug abuse within last 6 months
* Subjects who are otherwise considered to be ineligible for this study on investigators' judgment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in MDS UPDRS Part Ⅲ | From baseline (0d) after administration of the investigational product for 12 weeks
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. MDS-UPDRS Part III measures motor examination. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0(normal) to 4(severe).

SECONDARY OUTCOMES:
Change in the MDS UPDRS Part Ⅲ | After administration of the investigational product for 4 and 8 weeks
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. MDS-UPDRS Part III measures motor examination. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0(normal) to 4(severe).
Change in the MDS UPDRS Part Ⅰ | After administration of the investigational product for 4, 8, and 12 weeks
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I. MDS-UPDRS Part I measures non-motor experiences of daily living. Part I consists of 13 questions/evaluations, and each question is anchored with five response scale from 0(normal) to 4(severe).
Change in the MDS UPDRS Part Ⅱ | After administration of the investigational product for 4, 8, and 12 weeks
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II. MDS-UPDRS Part II measures motor experiences of daily living. Part II consists of 13 questions/evaluations, and each question is anchored with five response scale from 0(normal) to 4(severe).
Change in the MDS UPDRS Part Ⅰ+Part Ⅱ+Part Ⅲ | After administration of the investigational product for 4, 8, and 12 weeks
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I+II+III. MDS-UPDRS Part I measures non-motor experiences of daily living, Part II measures motor experiences of daily living and Part III measures motor examination. Part I and II each consists of 13 questions/evaluations and Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0(normal) to 4(severe).
Change in the Modified Hoehn and Yahr scale | After administration of the investigational product for 4, 8, and 12 weeks
  The Hoehn and Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress. The Hoehn and Yahr scale includes stages 1 through 5, with addition of stages 1.5 and 2.5 to help describe the intermediate course of the disease. The higher the score, the more severe the symptoms of Parkinson's disease progress.
Changes in each and total scores of K-NMSS | After administration of the investigational product for 4 and 12 weeks
  Korean version of Novel Non-Motor Symptoms Scale for Parkinson's Disease is 30-item scale containing nine dimensions: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems, attention/memory, gastrointestinal, urinary, sexual function and miscellany. Each symptoms are scored with severity (0=none, 1=mild, 2=moderate) and frequency (1=rarely, 2=often, 3=frequent, 4=very frequent). The final scores are calculated as severity score x frequency score. The higher the score, the severe the symptoms.
Change in the K-MoCA | After administration of the investigational product for 4 and 12 weeks
  The Montreal Cognitive Assessment (MoCA) is a screening assessment for detecting cognitive impairment. It is a 30-point test consisting of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points and a score of 26 or above is considered normal.
Changes in the summary index and total scores of the K-PDQ-39 | After administration of the investigational product for 4 and 12 weeks
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. Assessment is carried out across the 8 quality of life dimensions; activities of daily living, attention & working memory, cognition, communication, depression, functional mobility, quality of life, social relationships and social support. All items are scored from 0 (never) to 4 (always). Dimension score is then calculated by sum of scores of each item in the dimension divided by the maximum possible socre of all the items in the dimension, multiplied by 100. Lower dimension score reflects better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ok Nam Park, Study Director — Medihelpline Co., Ltd.
Locations (1):
- Yeouido St.Mary's Hospital, Yeongdeungpo-dong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided